CLINICAL TRIAL: NCT01049269
Title: Validation and Evaluation of a Portable Body Scanner for Determination of Obesity
Status: Completed | Type: Observational
Sponsor: University of Texas at Austin (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: R01DK081206; 5R21DK081206 (NIH)
Record Dates: First submitted 2010-01-13; First posted 2010-01-14 (Estimated); Last update posted 2015-06-25 (Estimated); Status verified 2007-01

CONDITIONS: Obesity
Keywords: Body Scanning; Body Fat; Body Volume; Obesity; No Conditions
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1:one group

SUMMARY:
The objective of this study is to validate a portable 3D human body measurement system which will improve approaches in obesity assessment.

DETAILED DESCRIPTION:
Obesity has become an epidemic in the United States. A new technique of three-dimensional (3 D) photonic scanning will be used to create and validate a portable instrument that rapidly assesses obesity in clinical and field settings. This new portable body scanner will be a safe and easy method to help determine the incidence and type of obesity.

ELIGIBILITY:
Inclusion Criteria:

* 18-60 years old
* BMI between 18.50 to 39.99 kg/m3
* Free of known diseases
* Hispanic and Not Hispanic or Latino Whites

Exclusion Criteria:

* Women who are pregnant, could be pregnant, or lactating

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Subject will be 18-60 years old, BMI 18.50 to 39.99 kg/m3, and free of known diseases, who are Hispanic and Not Hispanic or Latino Whites.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2007-01; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Body volume | 3 hours

SECONDARY OUTCOMES:
Validating body imaging as an indicator of central obesity | 3 hours

CONTACTS AND LOCATIONS:
Overall Officials: Jeanne H. Freeland-Graves, Ph.D., Principal Investigator — The University of Texas at Austin
Locations (1):
- The Uniersity of Texas at Austin, Austin, Texas, United States